CLINICAL TRIAL: NCT00076258
Title: Treatment With Exercise Augmentation for Depression (TREAD)
Brief Title: Adding Exercise to Antidepressant Medication Treatment for Depression
Acronym: TREAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Madhukar H. Trivedi, MD, Professor of Psychiatry, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU 092010-032; R01MH067692-01 (NIH)
Record Dates: First submitted 2004-01-16; First posted 2004-01-19 (Estimated); Results first posted 2016-12-07 (Estimated); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Depression
Keywords: Exercise therapy; Complementary Therapies
MeSH Terms: conditions — Depression | interventions — Selective Serotonin Reuptake Inhibitors; phosducin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SSRI+ LD (Experimental): A low dose aerobic exercise (LD) augmentation intervention to SSRI
  Interventions: Behavioral: SSRI + LD
- SSRI+ PHD (Experimental): A public health dose of aerobic exercise (PHD) augmentation intervention to SSRI
  Interventions: Behavioral: SSRI + PHD

INTERVENTIONS:
Behavioral: SSRI + LD — Eligible participants who have completed an adequate trial of SSRI monotherapy and all screening visits are randomly assigned to 24 weeks of SSRI augmentation with : a low dose of aerobic exercise (LD) or a public health dose of aerobic exercise (PHD). The acute phase of TREAD consists of the first 12 weeks of exercise augmentation intervention and includes: a) an individualized PHD- or LD aerobic exercise prescription; b) an empiricallybased behavioral intervention, including selfmonitoring tools and an interactive website, designed to maximize exercise adherence and minimize drop-out; and c) exercise instruction and supervised training sessions at The Cooper Institute (CI) as well as self-administered, home-based training sessions.
  Arms: SSRI+ LD
Behavioral: SSRI + PHD — Eligible participants who have completed an adequate trial of SSRI monotherapy and all screening visits are randomly assigned to 24 weeks of SSRI augmentation with : a low dose of aerobic exercise (LD) or a public health dose of aerobic exercise (PHD). The acute phase of TREAD consists of the first 12 weeks of exercise augmentation intervention and includes: a) an individualized PHD- or LD aerobic exercise prescription; b) an empiricallybased behavioral intervention, including selfmonitoring tools and an interactive website, designed to maximize exercise adherence and minimize drop-out; and c) exercise instruction and supervised training sessions at The Cooper Institute (CI) as well as self-administered, home-based training sessions.
  Arms: SSRI+ PHD

SUMMARY:
This study will assess the effectiveness of an exercise program in improving antidepressant medication treatment for individuals with major depressive disorder (MDD).

DETAILED DESCRIPTION:
Partial response to antidepressant treatment is common in people with MDD and is associated with significant morbidity and reduced quality of life. Pharmacological therapies have been used to augment the effect of antidepressants; however, such therapies are associated with a range of adverse effects. Studies indicate that exercise may be safe and effective in augmenting depression treatment. This study will determine whether exercise can complement selective serotonin reuptake inhibitor (SSRI) therapy in people with MDD who have residual symptoms of depression despite drug treatment.

Participants will be randomly assigned to either high frequency exercise or low frequency exercise for 12 weeks. Depression symptoms will be measured weekly. Quality of life and satisfaction with the study will also be measured. Depression scales and self-reports will be used to assess participants.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Major Depressive Disorder
* Score of 14 or higher on the Hamilton Depression Scale (HAM-D)
* 8 to 12 weeks of SSRI treatment, with at least 6 weeks at adequate doses
* Sedentary lifestyle
* Physically capable of exercise
* Body mass index (BMI) less than 40 kg/m2
* Willing and able to comply with study requirements

Exclusion Criteria:

* Significant cardiovascular disease or other medical conditions
* Uncontrolled hypertension
* Abnormal exercise stress test
* Hematologic disorders
* Comorbid disorders, including depression due to another comorbid condition, psychotic disorder, bipolar disorder, schizophrenia, schizoaffective disorder, eating disorder, or obsessive compulsive disorder (OCD)
* Alcohol and/or substance abuse in the past 6 months
* Hospitalization for mental illness within the past year
* High suicide risk
* Use of psychopharmacological or psychotherapeutic treatment other than SSRIs
* Failure to respond to two or more adequate pharmacological treatments during the current depressive episode
* Significantly elevated blood lipids
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2003-04; Primary Completion 2006-10 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhukar Trivedi, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center at Dallas, Dallas, Texas, United States

REFERENCES:
- [Background] Dunn AL, Trivedi MH, Kampert JB, Clark CG, Chambliss HO. The DOSE study: a clinical trial to examine efficacy and dose response of exercise as treatment for depression. Control Clin Trials. 2002 Oct;23(5):584-603. doi: 10.1016/s0197-2456(02)00226-x. PMID 12392873
- [Background] Dunn AL, Trivedi MH, O'Neal HA. Physical activity dose-response effects on outcomes of depression and anxiety. Med Sci Sports Exerc. 2001 Jun;33(6 Suppl):S587-97; discussion 609-10. doi: 10.1097/00005768-200106001-00027. PMID 11427783
- [Background] Crismon ML, Trivedi M, Pigott TA, Rush AJ, Hirschfeld RM, Kahn DA, DeBattista C, Nelson JC, Nierenberg AA, Sackeim HA, Thase ME. The Texas Medication Algorithm Project: report of the Texas Consensus Conference Panel on Medication Treatment of Major Depressive Disorder. J Clin Psychiatry. 1999 Mar;60(3):142-56. PMID 10192589
- [Background] Galper DI, Trivedi MH, Barlow CE, Dunn AL, Kampert JB. Inverse association between physical inactivity and mental health in men and women. Med Sci Sports Exerc. 2006 Jan;38(1):173-8. doi: 10.1249/01.mss.0000180883.32116.28. PMID 16394971
- [Background] Trivedi MH, Greer TL, Grannemann BD, Chambliss HO, Jordan AN. Exercise as an augmentation strategy for treatment of major depression. J Psychiatr Pract. 2006 Jul;12(4):205-13. doi: 10.1097/00131746-200607000-00002. PMID 16883145
- [Derived] Toups M, Carmody T, Greer T, Rethorst C, Grannemann B, Trivedi MH. Exercise is an effective treatment for positive valence symptoms in major depression. J Affect Disord. 2017 Feb;209:188-194. doi: 10.1016/j.jad.2016.08.058. Epub 2016 Oct 15. PMID 27936452
- [Derived] Suterwala AM, Rethorst CD, Carmody TJ, Greer TL, Grannemann BD, Jha M, Trivedi MH. Affect Following First Exercise Session as a Predictor of Treatment Response in Depression. J Clin Psychiatry. 2016 Aug;77(8):1036-42. doi: 10.4088/JCP.15m10104. PMID 27561137
- [Derived] Rethorst CD, Sunderajan P, Greer TL, Grannemann BD, Nakonezny PA, Carmody TJ, Trivedi MH. Does exercise improve self-reported sleep quality in non-remitted major depressive disorder? Psychol Med. 2013 Apr;43(4):699-709. doi: 10.1017/S0033291712001675. Epub 2012 Aug 29. PMID 23171815
- [Derived] Trivedi MH, Greer TL, Church TS, Carmody TJ, Grannemann BD, Galper DI, Dunn AL, Earnest CP, Sunderajan P, Henley SS, Blair SN. Exercise as an augmentation treatment for nonremitted major depressive disorder: a randomized, parallel dose comparison. J Clin Psychiatry. 2011 May;72(5):677-84. doi: 10.4088/JCP.10m06743. PMID 21658349

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SSRI+ LD | SSRI+ PHD
Started | 62 | 64
Completed | 61 | 61
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SSRI+ LD | SSRI+ PHD | Total
Number analyzed (Participants) | 61 | 61 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (9.4) | 45.6 (10.4) | 47.05 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 52 | 100
  Male | 13 | 9 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 60 | 61 | 121
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 5 | 9 | 14
  White | 54 | 51 | 105
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Hamilton Depression Rating Scale (17 item) [Mean (Standard Deviation); unit: units on a scale] — Hamilton Depression rating scale (17 item) is a clinical interview with scores that can range from 0-52. Higher scores indicate higher levels of depression symptoms.
  units on a scale | 18.1 (3.8) | 17.8 (3.8) | 17.9 (3.8)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Remission (Score of 12 or Less on Inventory for Depressive Symptomatology- Clinician-rated)
Description: The primary outcome measure- percentage of participants with remission (score of 12 or less on Inventory for Depressive Symptomatology- Clinician-rated). The change over time in probability of remission (IDS-C30 score ≤ 12) was compared between groups using a generalized linear mixed model (GLMM)41 as implemented in SAS (Proc Glimmix; SAS Institute Inc, Cary, North Carolina).
Time Frame: 12 weeks
Measure: Number; unit: percentage of participants in remission
Arm/Group | SSRI+ LD | SSRI+ PHD
Number analyzed (Participants) | 61 | 61
percentage of participants in remission | 18 | 18
Statistical Analysis 1: Comparison: SSRI+ LD vs SSRI+ PHD; Test type: Superiority or Other; p < 0.05, Generalized Linear Mixed Model; Both unadjusted and adjusted rates (for significant covariates) were reported; Remission rate = 29.5
Statistical Analysis 2: Comparison: SSRI+ LD vs SSRI+ PHD; For the covariate adjusted GLMM the remission rates were 15.5 for the LD and 28.3 for the PHD with a p < 0.06 and the NNT of 7.8 for the PHD versus the LD; Test type: Superiority or Other; p < 0.05, Generalized Linear Mixed Model; Remission Rate = 28.3

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | SSRI+ LD | SSRI+ PHD
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/64
Other Adverse Events (participants affected / at risk) | 62/62 | 64/64
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SSRI+ LD (N=62) | SSRI+ PHD (N=64)
Diarrhea, constipation, dry mouth and Nausea (Gastrointestinal disorders) | 52 (594) | 55 (598) — Specific adverse event terms are unknown because adverse events were only collected with regard to the affected organ system.
Palpitation, dizzy and chest pain (Cardiac disorders) | 29 (188) | 33 (143) — Specific adverse event terms are unknown because adverse events were only collected with regard to the affected organ system.
Rash, perspiration, itching and dry skin (Skin and subcutaneous tissue disorders) | 51 (600) | 49 (620) — Specific adverse event terms are unknown because adverse events were only collected with regard to the affected organ system.
Headache, tremors, coordination and dizzy (Nervous system disorders) | 56 (604) | 56 (515) — Specific adverse event terms are unknown because adverse events were only collected with regard to the affected organ system.
Blurred vision /ears ringing (Eye disorders) | 36 (207) | 25 (288) — Specific adverse event terms are unknown because adverse events were only collected with regard to the affected organ system.
Difficult urination, painful urination,frequent urination and irregular menstruation (Renal and urinary disorders) | 28 (186) | 28 (125) — Specific adverse event terms are unknown because adverse events were only collected with regard to the affected organ system.
Difficulty sleeping, sleeps too much (Psychiatric disorders) | 58 (621) | 61 (532) — Specific adverse event terms are unknown because adverse events were only collected with regard to the affected organ system.
loss of desire, trouble orgasm and trouble erections (Reproductive system and breast disorders) | 50 (521) | 40 (377) — Specific adverse event terms are unknown because adverse events were only collected with regard to the affected organ system.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No